CLINICAL TRIAL: NCT01171690
Title: Pilot Study of Teriparatide for Postsurgical Hypoparathyroidism
Brief Title: Teriparatide for Postsurgical Hypoparathyroidism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding problems
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marius Stan, Assistant Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-000901
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Hypoparathyroidism Post-surgical
Keywords: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Teriparatide (Experimental): The dose of teriparatide will be 20 mcg twice daily for the first week and 20 mcg daily for the second week. If hypocalcemia recurs after 2nd week, teriparatide will be continued for a 3rd week and then discontinued.
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — The dose of teriparatide will be 20 mcg twice daily for the first week and 20 mcg daily for the second week. If hypocalcemia recurs after 2nd week, teriparatide will be continued for a 3rd week and then discontinued.
  Other Names: Forteo

SUMMARY:
This study evaluated the effects of teriparatide (Forteo) on low calcium levels in the setting of thyroid surgery associated with low parathyroid hormone. The hypothesis was that teriparatide ( Forteo) would shorten the length of hospitalization post thyroidectomy in patients with symptomatic hypoparathyroidism.

DETAILED DESCRIPTION:
Transient hypoparathyroidism with hypocalcemia occurs in up to 20 % of patients after surgery for thyroid cancer, multinodular goiter or Graves' disease and is severe in around 3 to 18% of cases. Severe hypocalcemia significantly lengthens their hospital stay. This study will evaluate the effects of teriparatide (synthetic parathyroid hormone, brand name Forteo) on low calcium levels in the setting of thyroid surgery associated with low parathyroid hormone.

This was a feasibility open-label, single-arm trial with historical matched controls with a planned enrollment of 15 patients with severe, symptomatic hypocalcemia that would be treated with teriparatide for a maximum duration of 3 weeks and compared the active subjects with 30 gender and age matched controls.

Therapy for hypocalcemia continued in accordance with current practice. The decision for discharge, as far as calcium is concerned, was to be reached when calcium level was > 7.5 mg/dL and increased x 2 over 12 hours in an asymptomatic patient with stable therapy and no need for IV calcium in the last 24 hours. Subjects were followed by phone and with blood tests 2 days after discharge and 9, 17 and 25 days after initiation of teriparatide. They were off teriparatide for 24 hours prior to testing on days 9, 17 and 25.

If hypocalcemia recurred after 2nd week, teriparatide was continued for a 3rd week and then discontinued. If hypocalcemia recurred again current standard therapy for hypoparathyroidism was continued off teriparatide.

ELIGIBILITY:
Inclusion criteria:

* Patients post bilateral thyroid bed surgery (cancer, Graves disease, multinodular goiter)
* Symptomatic hypocalcemia
* Total calcium < 8 mg/dL persisting after 24 hours of therapy with calcitriol (minimum 0.25 mcg twice a day) and calcium supplementation (minimum 1.5 grams of elemental calcium per day)
* Parathyroid hormone (PTH) level below low end of normal range

Exclusion criteria (all subjects):

* Renal failure
* Any prior parathyroid pathology
* Pre-existing hypercalcemia
* Metabolic bone diseases other than osteoporosis
* Pagets disease

Exclusion criteria (active treatment subjects only):

* Ongoing therapy with Forteo for osteoporosis
* Active non-thyroidal malignancy or suspicion of residual thyroid malignancy
* History of skeletal malignancies, primary or metastatic
* Pregnancy
* Active or recent urolithiasis
* Digitalis therapy
* Patients at increased baseline risk for osteosarcoma, i.e., family history of osteosarcoma or prior radiation therapy involving the skeleton
* Pediatric populations
* Unexplained elevations of alkaline phosphatase

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Stan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited between 1/1/2010 and 1/12/2013; all patients were recruited at Mayo Hospitals in Rochester, Minnesota, USA. The controls were recruited from the pool of patients with similar degree of hypoparathyroidism postoperatively but previously to the initiation of the trial.
Groups:
- Control: These are patients with similar degree of hypocalcemia that were treated per standard of care for hypoparathyroidism and did not receive teriparatide. They were all hospitalized at the time of hypocalcemia and were matched by age and gender with the intervention group.
Period: Overall Study
Arm/Group | Teriparatide | Control
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with severe and symptomatic hypocalcemia within the first 24 hours postoperatively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Control | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [31 to 53] | 40 [32 to 57] | 41 [31 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Hospital length of stay from initiation of therapy with calcium and calcitriol to "ready to discharge" from a calcium perspective (calcium level > 7.5 mg/dL and increasing x 2 over 12 hours in an asymptomatic patient with stable therapy and no need for intravenous (IV) calcium in last 24 hours).
Time Frame: Approximately 7 days after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 5 | 5
days | 1.1 (0.4) | 2.4 (1.1)
Statistical Analysis 1: Comparison: Teriparatide vs Control; Matched pairs; Test type: Superiority or Other; p = 0.01, Matched pairs t test

2. Secondary Outcome: Safety Analysis
Description: Arms were compared for total number of adverse events, including severe and serious adverse events.
Time Frame: Approximately 90 days after surgery
Measure: Number; unit: events
Arm/Group | Teriparatide | Control
Number analyzed (Participants) | 5 | 5
events | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months after starting the intervention
Groups:
- Teriparatide: The dose of teriparatide will be 20 mcg twice daily for the first week and 20 mcg daily for the second week. If hypocalcemia recurs after 2nd week, teriparatide will be continued for a 3rd week and then discontinued.
  There were no adverse events related to the use of teriparatide.
Arm/Group | Teriparatide | Control
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes